CLINICAL TRIAL: NCT05760352
Title: Comparison of Multiple Methods of Exercise Training for Accessing Maximal Oxygen Consumption, Skeletal Muscle Oxygen Saturation, and Cardiopulmonary Outcomes in Patients With Chronic Respiratory Disease
Brief Title: Comparison of Multiple Exercise Trainings in Chronic Respiratory Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FJUH111193
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Chronic Pulmonary Disease
Keywords: Pulmonary rehabilitation; Eccentric cycling exercise; Helmet ventilation; Chronic respiratory disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Self-paced exercise
- Intervention Group: eccentric cycling exercise (Experimental): Received eccentric cycling exercise
  Interventions: Device: Eccentric bike
- Intervention Group: eccentric cycling exercise with helmet ventilation (Experimental): Eccentric cycling exercise combined with helmet ventilation
  Interventions: Device: Eccentric bike; Device: Helmet ventilation

INTERVENTIONS:
Device: Eccentric bike — Received eccentric cycling exercise
  Arms: Intervention Group: eccentric cycling exercise; Intervention Group: eccentric cycling exercise with helmet ventilation
Device: Helmet ventilation — Using helmet ventilation during eccentric cycling exercise
  Arms: Intervention Group: eccentric cycling exercise with helmet ventilation

SUMMARY:
The present study aims to investigate the effect of different exercise training in patients with chronic respiratory disease.

DETAILED DESCRIPTION:
Background： Chronic respiratory and chronic obstructive pulmonary disease is the one of the major causes of global morbidity and mortality. Patients with chronic respiratory disease often experience exercise limitation and physical inactivity due to muscular weakness and severe dyspnea. Symptoms of COPD may contribute to activity restriction, deconditioning, and exercise intolerance. Pulmonary rehabilitation has been demonstrated to improve clinical outcomes and exercise capacity in patients with chronic respiratory disease. However, the optimal exercise training modality is remaining unclear.

Study Design： This is a one-year, single-centre, prospective randomized controlled trial

Methods： The investigators expected a total of 60 participants were be enrolled, then randomly assigned into three groups (control group, experimental-1, and experimental-2). All participants will receive a graded exercise test, then followed a 9-weeks of exercise training. After 9-weeks of exercise training, the maximal oxygen consumption will be analyzed as a primary outcome of this study. Physiological parameters, hemodynamic outcome, respiratory function, and strength of lower limb muscle will be recorded.

Effect： After 9 weeks' exercise training, VO2 will significantly improve in eccentric cycling exercise groups, furthermore, heart rate and perceived exertion will be lower in the eccentric cycling exercise combined with helmet ventilation.

Key words： Pulmonary rehabilitation; eccentric cycling exercise; helmet ventilation; chronic respiratory disease

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 80 years
* Diagnosed with chronic respiratory diseases
* Having undergone pulmonary rehabilitation for more than 3 months

Exclusion Criteria:

* Existing of tracheostomy
* Those who use oxygen therapy or ventilator at home
* Severe left heart failure (NYHA III-IV)
* Neuromuscular disease
* Acute exacerbation within the past three months
* Those who are unable to cooperate with the cardiopulmonary exercise test

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Peak % of oxygen consumption | 9 weeks
  To observe the maximum exercise performance

SECONDARY OUTCOMES:
Heart rate, b/m | 9 weeks
  Cardiac hemodynamic parameter
Respiratory rate, b/m | 9 weeks
  Pulmonary parameter
Mean arterial blood pressure, mmHg | 9 weeks
  Cardiac hemodynamic parameter
FEV1/FVC, % | 9 weeks
  Pulmonary function
Saturation of Peripheral Oxygen(SpO2), % | 9 weeks
  Blood oxygenation

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No